CLINICAL TRIAL: NCT02456246
Title: Piloting the Feasibility of FLT-PET/CT Non-Small Cell Lung Cancer Managed With SBRT
Acronym: SBRT FLT-PET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UHN REB 15-8972-CE
Record Dates: First submitted 2015-05-26; First posted 2015-05-28 (Estimated); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Non Small Cell Lung Cancer (NSCLC)
Keywords: Stereotactive Body Radiation Therapy (SBRT); Lung Fibrosis; FLT-PET; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Pulmonary Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FLT-PET (Experimental): 1. Cohort 1: Patients in this cohort would be treatment naïve and will be planned for SBRT treatment according to established institutional practices. FLT-PET in this subgroup will be performed before radiation therapy.
  2. Cohort 2: Patients who have had SBRT and demonstrate typical or stable lung fibrosis on follow up CT
  3. Cohort 3: Patients who have had SBRT and demonstrate findings suspicious for recurrence on follow up CT or who have biopsy demonstrating disease recurrence.
  Interventions: Procedure: FLT-PET

INTERVENTIONS:
Procedure: FLT-PET — Positron emission tomography scan using the 18f-FLT (3'deoxy-3'-fluorothymidine) tracer

SUMMARY:
Stereotactic body radiotherapy (SBRT) has emerged as one of the leading curative method for early stage non-small cell lung cancer (NSCLC). However, assessing the status of the disease during post-SBRT follow up presents a challenge. Currently, chest Computed Tomography (CT) is the main technique to detect whether cancer has come back, but this method has demonstrated poor accuracy and reliability in determining if the observed post-operative lung changes are benign or malignant.

Positron-emission tomography (PET) is an imaging technique that uses special radioactive tracers to cell growth. The use of PET scans with a tracer that target the pathways of DNA synthesis may be more accurate than CT for detecting if the cancer has come or not.

The purpose of this study is to see if a PET radiotracer called 18F-FLT (3'-deoxy-3'-fluorothymidine) can identify cancer recurrences accurately compared to regular CT scans.

DETAILED DESCRIPTION:
Stereotactic body radiotherapy (SBRT) has demonstrated an impressive 3-year control rate of higher than 90% for early stage NSCLC, leading to increased use of this technique as a curative method for lung cancer treatment. With growing clinical experience with this technique, post-SBRT follow up has received more attention. Follow up after SBRT is done primarily by thorax CT, which is affected by radiation-induced radiographic lung changes that can resemble or obscure local recurrence.

FLT (3'-deoxy-3'-fluorothymidine) is a thymidine analogue which is non-toxic in tracer doses, and can be labeled with 18F. FLT-PET is a type of imaging (similar concept to the widely used 18-FDG PET-CT) that is based on integration of thymidine into DNA for assessment of proliferation. Conceptually, increased DNA synthesis is correlated to tumor aggressiveness and response to therapy, more so than glucose utilization - as in FDG-PET could be.

The purpose of this study is therefore to see what added information the use of FTL-PET can provide in distinguishing between changes in the lung that occur as a result of treatment that are not cancerous and those that are due to recurrence or progressive disease.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Must have been treated at or plan to be treated at Princess Margaret Cancer Centre with SBRT for an early-stage NSCLC (T1N0M0; T2N0M0; or T3N0M0 chest wall primary tumours only) and are either:

   1. Prior to treatment with lung SBRT (for Cohort 1)
   2. Have radiographic findings on that are felt to be related to fibrosis at any time point following lung SBRT
   3. Have radiographic findings on CT that are suspicious for recurrence at any time point following lung SBRT
3. Ability to provide written informed consent to participate in the study

Exclusion Criteria:

1. Previous systemic therapy
2. Previous thoracic radiotherapy(excluding the index lung SBRT treatment)
3. Active malignancy other than lung cancer
4. Unable to remain supine for more than 30 minutes
5. If taking the drug Antabuse
6. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2023-02-24 (Actual); Study Completion 2023-02-24 (Actual)

PRIMARY OUTCOMES:
To report the SUVmax for the three cohorts | 1 year

SECONDARY OUTCOMES:
To compare FLT uptake in 4D (respiratory sorted) versus free breathing FLT-PET scans | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Meredith Giuliani, MD, Principal Investigator — UHN
Locations (1):
- University Health Network, Toronto, Ontario, Canada